CLINICAL TRIAL: NCT01187394
Title: Plasma Utilization Following Cardiac Surgery
Acronym: PUCS
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Blood Services (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2009769 01
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Blood Component Transfusion; Cardiac Surgical Procedures
Keywords: Frozen Plasma; Fresh Frozen Plasma; Cardiac Surgery; Bleeding; Knowledge Translation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In Canada, 218,000 units of fresh frozen plasma and frozen plasma were transfused in 2005.Cardiac surgery patients are the largest recipient group for FP transfusions. Despite this, no studies have characterized the use of FP in relation to coagulation test abnormalities or bleeding, or how these and other clinical determinants influence the decision to transfuse FP. Furthermore, no studies have evaluated the effectiveness of FP transfusions in correcting laboratory abnormalities or treating bleeding in cardiac surgery.

Given the varied use of FP transfusions in cardiac surgery, further studies are essential.In order to improve current utilization of FP, current use must be understood, and the relationship between FP transfusions and the clinical factors that affect the decision to transfuse FP.

DETAILED DESCRIPTION:
This study will examine (1) the utilization pattern in the use of FP transfusions, (2) the clinical determinants influencing physician's decision to transfuse and blood loss and (3) coagulation tests in individual cardiac surgery patients. Through greater understanding of the current use of FP in cardiovascular surgery, we can improve its utilization and reduce unnecessary and harmful exposure to blood products.

Objectives: We will describe the incidence and clinical determinants of FP transfusions in cardiac surgery. Secondarily, we will evaluate the relationships between the utilization of FP transfusions and (1) blood loss and (2) coagulation test results.

Methods: All FP transfusions given to cardiac surgery patients intra and postoperatively in the intensive care unit will be reviewed. At the time of the transfusion (intraop) or request (postop) for FP all physicians will complete a short questionnaire evaluating the clinical factors influencing their decision to transfuse. For a sample of postoperative patients with elevated an INR who are not transfused FP, we will have physicians complete a similar short questionnaire evaluating the same clinical factors. Charts of all cardiac surgery patients will be reviewed to capture baseline, intraoperative and postoperative data including demographics, transfusions, blood loss and laboratory results. Charts of patients with INR > 1.2 and/or receiving FP will be reviewed in detail to collect baseline data, intraoperative data, and detailed post operative data including FP transfusions, other blood transfusions, blood loss, lab and coagulation results, and adverse transfusion reactions. Data will collected for duration of stay in intensive care.

Outcomes: The primary outcomes are the (i) the proportion of patients transfused FP and the dose of FP transfused and (2) the importance the clinical determinants influencing the decision to transfuse FP. Secondary outcomes include measures of blood loss (mediastinal chest tube blood loss, change in hemoglobin and number of red blood cell transfusions), changes in coagulation tests results (INR, PTT), the frequency of adverse transfusion reactions, length of ICU and hospital stay, and mortality.

Analysis: The primary analysis will be a descriptive analysis of FP transfusions and the clinical determinants influencing the decision to transfuse FP. A multivariable logistic regression analysis will be performed to examine the variables associated with FP utilization including the postoperative IN, hemoglobin, red cell transfusions and mediastinal chest tube loss in patients transfused FP. The correlation between the physician reported clinical determinants for FP transfusions and blood loss and coagulation test results will be examined by Spearman and Pearson correlations as appropriate , and multiple logistic regression. For the analysis of secondary outcomes, the mean change in blood loss and coagulation test results following FP transfusion will be calculated, and a multivariable regression analysis will be performed to examine the relationship between blood loss, FP transfusions and changes in the INR.

ELIGIBILITY:
Inclusion Criteria:

*All subjects undergoing Cardiopulmonary Bypass surgery

More detailed Data Collection for subjects:

* who either receive at least one Frozen Plasma Transfusion or
* who have an INR > 1.2 in the 72 hours following surgery and
* are admitted to an intensive care unit.

Exclusion Criteria:

* No subjects undergoing cardiopulmonary bypass surgery will be excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at six 6 Canadian Centres
Sampling Method: Non-Probability Sample
Enrollment: 970 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Frozen Plasma Transfusion | 1 month
  For FP Transfusions, we will determine the proportion of patients transfused FP for (a) all cardiac surgery patients, (b) for patients with an INR> 1.2, (c) for patients with an INR > 1.5 and (d) for patients with no recent coagulation tests available. We will also determine the number of units and volume (mL/kg) for each transfusion order and the total number of units and volume (mL/kg) transfused in addition to the timing of all units transfused in the first 72 hours after cardiac surgery.

SECONDARY OUTCOMES:
Clinical determinants influencing the decision to transfuse | 1 month
  We will examine seven clinical determinants that may influence the decision to transfuse: (1) change in hemoglobin, (2) ongoing chest tube blood loss, (3) potential future blood loss, (4) INR/PT results, (5) aPTT results, (6) hemodynamic instability, (7) hemodilution. We will capture the importance of these factors using a visual analog scale. The same seven clinical determinants will be examined for patients with an elevated INR who are not transfused FP

CONTACTS AND LOCATIONS:
Overall Officials: Alan T Tinmouth, MD MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada